CLINICAL TRIAL: NCT07285252
Title: ENDURE- Evaluating Non-Invasive Haptics During Extreme Exercise
Brief Title: Evaluating Non-Invasive Haptics During Extreme Exercise
Acronym: ENDURE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: SuperPatch Limited LLC (Industry)
Collaborators: Clarity Science LLC (Unknown); The Altitude Centre (Unknown); Vichag Healthcare Research (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ENDURE-001
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-12

CONDITIONS: VO2max; Lactate Threshold; Lactate
Keywords: VO2 max; lactate threshold; lactate

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomised, double-blinded, parallel-group internal pilot study evaluating the acceptability, safety, recruitment processes, data-collection procedures, and preliminary performance signals of the SuperPatch VICTORY vibrotactile patch in recreational-competitive runners. The Study was designed to inform a future fully-powered interventional study. The study follows the CONSORT Extension for Pilot and Feasibility Trials. The study involves comparison of data from two parallel groups: (1) an active intervention group using SuperPatch VICTORY Patch (intervention) versus (2) a placebo group using a visually identical patch lacking the vibrotactile neurosensory pattern. Participants will be followed for four weeks with lab-based assessments at baseline (Week 0), Week 2, and Week 4.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATMENT (Active Comparator): Victory Patch
  Interventions: Device: Victory Patch with Haptic Vibrotactile Trigger Technology
- CONTROL (Placebo Comparator): Sham Comparator
  Interventions: Device: Sham patch

INTERVENTIONS:
Device: Victory Patch with Haptic Vibrotactile Trigger Technology — Active Patch with Haptic Vibrotactile Trigger Technology
  Arms: TREATMENT
Device: Sham patch — Sham/Placebo Patch without Haptic Vibrotactile Trigger Technology
  Arms: CONTROL

SUMMARY:
This study aims to compare determinants of endurance performance between participants wearing an active patch with haptic vibrotactile trigger technology (VTT) versus a placebo patch without VTT among recreational to competitive runners over a 4-week training period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and over, that participate in recreational to competitive distance running (>2 structured runs per week), that were able to complete maximal treadmill exercise safely and were able to attend three laboratory visits were invited to participate.

Exclusion Criteria:

* Adults with a contraindications to high-intensity treadmill exercise, cardiovascular, metabolic, or musculoskeletal conditions limiting participation, reported use of performance-enhancing drugs, pregnancy, known allergy to adhesives, or current use of neuromodulatory or haptic devices

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in VO2 Max | 2-weeks and 4-weeks after baseline assessment
  Change in VO₂max (mL/kg-¹/min-¹, calculated as a 30-second rolling average)

SECONDARY OUTCOMES:
Change in Lactate-threshold running speed | 2-weeks and 4-weeks after baseline assessment
  Measurement of Lactate-threshold running speed using capillary sampling (LT, km/h-¹), determined using a DmodMax algorithm on lactate-speed curves [15], (2) serum lactate level at threshold (mmol·L-¹).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sakr, DO, Principal Investigator — University of Arizona
Locations (1):
- The Altitude Centre, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon Initiation of the Study
Access Criteria: Current Study Investigators and associated Research Staff